CLINICAL TRIAL: NCT07272616
Title: A Prospective Comparative Study of a Novel Gadolinium-Weighted MRI Sequence Versus Conventional T1-Weighted Imaging for the Detection of Brain Metastases
Brief Title: Detection of Brain Metastases Using a Novel Gadolinium-Weighted MRI Sequence: A Prospective Comparison
Acronym: GDW
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K2025-9115
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Suspected or Known Brain Metastases: Participants undergoing clinically indicated brain MRI with gadolinium contrast who will receive both conventional T1-weighted imaging and the novel gadolinium-weighted MRI sequence during the same scan session. The purpose is to compare lesion detection and conspicuity between the two sequences.
  Interventions: Diagnostic Test: Novel Gadolinium-Weighted MRI Sequence

INTERVENTIONS:
Diagnostic Test: Novel Gadolinium-Weighted MRI Sequence — A post-contrast MRI sequence incorporating magnetization transfer (MT) preparation and flow-nulling with motion-sensitized driven equilibrium (MSDE). The sequence is optimized to suppress background tissue and vascular signal while enhancing the visibility of gadolinium-enhancing brain metastases. It is compared to conventional T1-weighted imaging in the same exam session.

SUMMARY:
This study will evaluate a new type of MRI sequence designed to improve the visibility of brain metastases after gadolinium contrast injection. The purpose is to determine whether this novel "gadolinium-weighted" imaging method can detect more or smaller tumors than standard MRI techniques. Participants will undergo a routine brain MRI with contrast, followed by an additional scan using the new method. The goal is to improve diagnostic accuracy without increasing the contrast dose or scan time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for clinical brain MRI with gadolinium contrast
* Known or suspected brain metastases
* Able to provide informed consent
* Able to lie still for the duration of the MRI examination

Exclusion Criteria:

* Contraindications to MRI
* Known allergy or contraindication to gadolinium-based contrast agents
* Renal impairment (eGFR < 30 mL/min/1.73m²)
* Pregnant or breastfeeding
* Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for clinical brain MRI with contrast at a university hospital radiology department in Sweden. Participants will be adults with known or suspected brain metastases undergoing routine post-gadolinium imaging as part of their diagnostic work-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Number of Detected Gadolinium-Enhancing Brain Metastases Between the Novel Gadolinium-Weighted MRI Sequence and Conventional T1-Weighted Imaging | At the time of gadolinium-enhanced MRI, during a single imaging session (within 1 hour of contrast administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No